CLINICAL TRIAL: NCT02077088
Title: Double Blind, Randomised Study on the Effect of Prebiotics on Incidence of Atopic Manifestations in Infants
Brief Title: Effect of Galactooligosaccharides on Incidence of Atopic Manifestations in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humana Co.Ltd. (Industry)
Collaborators: Vitkovice Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1.090
Record Dates: First submitted 2014-01-02; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Atopic Dermatitis
Keywords: interventional; doubleblind; randomised; pediatric; prebiotic; atopic; dermatitis; infant
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — 4'-galactooligosaccharide; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galactooligosaccharides (Experimental): addition of 0,5g galactooligosaccharides to HA (hypoallergenic) starter formula
  Interventions: Other: galactooligosaccharide
- Only HA formula (No Intervention): only standard HA starter formula

INTERVENTIONS:
Other: galactooligosaccharide — addition of food grade GRAS (Generally Regarded As Safe) galactooligosaccharides
  Other Names: GOS; prebiotics
  Arms: Galactooligosaccharides

SUMMARY:
Addition of prebiotic galactooligosaccharides to hypoallergenic starter formula would lead to decreased allergic (atopic) symptoms in nonbreastfed infants with a positive history of allergy in family

ELIGIBILITY:
Inclusion Criteria:

* nonbreastfed eutrophic infants of corresponding gestational age
* presence of a positive family allergic anamnesis in parents or siblings (atopic eczema, allergic rhinitis or bronchial asthma)

Exclusion Criteria:

* children with serious disease,
* breastfed children
* children fed another formula then the ones used

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
SCORAD (SCORing Atopic Dermatitis score) assessment of atopy | at 6 months of age
  objective evaluation of atopic symptoms

SECONDARY OUTCOMES:
anthropometric parameters (height, weight) | at 6 months of age

OTHER OUTCOMES:
incidence of febrile episodes | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bozensky, MD, Principal Investigator — Vitkovice Hospital, Ostrava, Czech Republic
Locations (1):
- Vitkovice Hospital, Ostrava-Vitkovice, Czechia

REFERENCES:
- [Derived] Bozensky J, Hill M, Zelenka R, Skyba T. Prebiotics Do Not Influence the Severity of Atopic Dermatitis in Infants: A Randomised Controlled Trial. PLoS One. 2015 Nov 16;10(11):e0142897. doi: 10.1371/journal.pone.0142897. eCollection 2015. PMID 26571488